CLINICAL TRIAL: NCT02817022
Title: Evaluation of the Effect of Application of Developmentally Supportive Care on Neurobehavioral Outcome of Preterm Very Low Birth Weight Neonates
Brief Title: Developmentally Supportive Care on Neurobehavioral Outcome of Preterm Very Low Birth Weight Neonates
Acronym: DSC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lady Hardinge Medical College (Other Government)
Responsible Party: Principal Investigator, DR. VIKRAM DATTA, professor, Lady Hardinge Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Developmental supportive care
Record Dates: First submitted 2016-04-29; First posted 2016-06-29 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Very Low Birth Weight Baby
Keywords: Developmentally Supportive Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- developmentally supportive care (Other): enrolled neonates will be provided routine supportive care as per existing NICU protocols. This will be carried out in the initial 6 months (0-180 days) of study commencement. This group will serve as control group (group A). During subsequent 6 months (181-360 days) of the study period, enrolled neonates fulfilling the inclusion criteria will be provided routine supportive care and the components of developmentally supportive care(DSC). DSC components will be strictly emphasized on protected sleep, pain and stress assessment and management, activities of daily living (positioning, feeding and skin care), the healing environment. This group will be designated as group B
  Interventions: Other: developmentally supportive care

INTERVENTIONS:
Other: developmentally supportive care — DSC components will be strictly emphasized on protected sleep, pain and stress assessment and management, activities of daily living (positioning, feeding and skin care), the healing environment

SUMMARY:
Enrolled neonates will be provided routine supportive care as per existing neonatal intensive care unit (NICU)protocols. This will be carried out in the initial 6 months (0-180 days) of study commencement. This group will serve as control group (group A). During subsequent 6 months (181-360 days) of the study period, enrolled neonates fulfilling the inclusion criteria will be provided routine supportive care and the components of developmentally supportive care (DSC).

DETAILED DESCRIPTION:
Enrolled neonates will be provided routine supportive care as per existing NICU protocols. This will be carried out in the initial 6 months (0-180 days) of study commencement. This group will serve as control group (group A). During subsequent 6 months (181-360 days) of the study period, enrolled neonates fulfilling the inclusion criteria will be provided routine supportive care and the components of developmentally supportive care (DSC). DSC components will be strictly emphasized on protected sleep, pain and stress assessment and management, activities of daily living (positioning, feeding and skin care), the healing environment. This group will be designated as group B. Both the groups will receive appropriate management for their morbidities as per existing NICU protocols. Both the groups will be followed up till 37 weeks of gestation where in their neurobehavioral assessment will be performed using Neurobehavioural assessment of preterm infants score.

In both the groups all the baseline data regarding antenatal factors will be recorded in a predesigned proforma such as age, gravid, Gestational age, Chorioamnionitis, Prenatal steroids, Multiple pregnancy, maternal comorbidities (preeclampsia, gestational diabetes mellitus), mode of delivery etc.

ELIGIBILITY:
Inclusion Criteria:

* All stable preterm very low birth weight babies not on invasive mechanical ventilation
* Hemodynamically stable
* Parental consent

Exclusion Criteria:

* Babies with major congenital anomalies
* Asphyxia (Apgar score <3 at 5mins).
* Acute bilirubin encephalopathy
* Hypoglycemia at enrollment
* Clinical Chorioamnionitis(fever > 100.4 ◦ f , uterine fundal tenderness, maternal tachycardia (>100/min), fetal tachycardia (>160/min) and purulent or foul amniotic fluid )
* History of birth trauma

Ages: 1 Day to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Neurobehavioral outcome Of the Preterm Very low birth weight babies | 18 months
  Neurobehavioural outcome will be measured by NAPI at 37 weeks of corrected gestational age.

SECONDARY OUTCOMES:
Time to achieve full feeds @150ml/kg | 18 months
  Time to achieve full feed @150 ml/kg/day will be measured in days.
Length of hospital stay | 18 months
  will be measured in days

OTHER OUTCOMES:
Number of apneic episodes during hospital stay | 18 months
  will be measured as per standard definition of neonatal apnea and expressed as numbers.
IVH Grade 2 or more | 18 months
  will be measured using bedside cranial sonogram and classified using Volpe's classification.
BPD | 18 months
  Presence or absence will be noted and mentioned as yes or no.
NEC Stage 2 or more | 18 months
  Will be staged using Bells staging .
ROP (any stage) | 18 months
  Will be graded using standard classification .

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - Lady Hardinge Medical College, New Delhi, National Capital Territory of Delhi
  - Lady Hardinge Medical College,New Delhi, Delhi

IPD SHARING:
Plan to Share IPD: Undecided